CLINICAL TRIAL: NCT03884205
Title: GDPE/CEOPE Compared With CEOPE as the First-line Therapy for Newly Diagnosed Patients With Peripheral T-Cell Lymphoma
Brief Title: GDPE/CEOPE Compared With CEOPE for Newly Diagnosed Patients With PTCL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Wang Xin, Department Director, Shandong Provincial Hospital
Other Study IDs: Gemcitabine-PTCL
Record Dates: First submitted 2019-03-16; First posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: PTCL; Gemcitabine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- test group: patients with PTCL who receive GDPE/CEOPE as the first-line therapy strategy
- control group: patients with PTCL who receive CEOPE as the first-line therapy strategy

SUMMARY:
Peripheral T-cell Lymphoma (PTCL) is a heterogenic malignancy with poor outcome. There is no standardized treatment protocol for this kind of lymphoma. So, clinical trials are encouraged by National Comprehensive Cancer Network (NCCN) for those patients. Former studies confirmed that GDP (Gemcitabine, Dexamethasone, and Cis-platinum) is superior with CHOP (Cyclophosphamide, Adriamycin, Vincristine, and Prednisone). Combination with etoposide can improve the outcome of some patients with high risk factors. The aim of our study is to compare the response and survival rate of GDPE/CEOPE (gemcitabine, cis-platinum, etoposide, and dexamethasone/cyclophosphamide, vincristine, pharmorubicin, etoposide, and prednisone) with those of CEOPE regimen, looking forward to its superiority in efficacy and safety for the newly diagnosed adult patients with PTCL.

DETAILED DESCRIPTION:
Peripheral T-cell Lymphoma (PTCL) is a heterogenic malignancy with poor outcome. Five-year PFS (progression-free survival) and OS (overall survival) for these patients received classic CHOP regimen is less than 30%. High-dose intensive chemotherapy doesn't demonstrate better response. At present, there is no standardized treatment protocol for this kind of lymphoma. So, clinical trials are encouraged by NCCN for those patients.

For the less efficacy of CHOP or CHOP-like regimen, multi-drug combination strategy has been the therapy tendency in PTCL. Zhang et al, reported that GDP compared with CHOP as the therapy strategy for PTCL-NOS (Not Otherwise Specified). The response rate was 78.57% in GDP group and 60.00% in CHOP group, respectively. DFS (disease-free survival) was 9.79 and 4.2 months in above two groups. They concluded that GDP is superior to CHOP. The main side-effect of two regimens is hematological toxicity. Combination with etoposide can improve the outcome of some patients with high risk factors. Furthermore, high-dose combined with ASCT (autologous stem cell transplantation) has been the first-line therapy for PTCL. Some refractory/relapsed patients with PTCL will benefit from allogeneic bone marrow transplantation. However, about 30% patients with PTCL have no chance to receive ASCT for multiple reasons. So, it is urgent to explore new combination-therapy regimen to improve the outcome for patients with PTCL.

The aim of our study is to compare the response and survival rate of GDPE/CEOPE (gemcitabine, cis-platinum, etoposide, and dexamethasone/cyclophosphamide, vincristine, pharmorubicin, etoposide, and prednisone) with those of CEOPE (/cyclophosphamide, vincristine, pharmorubicin, etoposide, and prednisone ) regimen, looking forward to its superiority in efficacy and safety for the newly diagnosed adult patients with PTCL.

ELIGIBILITY:
Inclusion Criteria:

* Peripheral T Cell Lymphoma, Not Otherwise Specified
* Angioimmunoblastic T Cell Lymphoma
* ALK-negative Anaplastic Large Cell Lymphoma
* Enteropathy Associated T Cell Lymphoma
* Subcutaneous Panniculitis Like T Cell Lymphoma
* Acute T-cell Leukemia/Lymphoma

Exclusion Criteria:

* woman in pregnancy or lactation
* allergic to any intervention drug
* unsuitable to the study due to severe complication
* enrolled to other study during the past 6 months
* NK/T lymphoma ALK-positive Anaplastic Large Cell Lymphoma

Ages: 16 Years to 75 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Newly Diagnosed Patients with Peripheral T-cell Lymphoma (PTCL)
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
RR | 1 year
  Response Rate (including complete response & partial response)

SECONDARY OUTCOMES:
PFS | 1 year
  progression free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Yujie MS JIANG, Jinan, SD, China

IPD SHARING:
Plan to Share IPD: No